CLINICAL TRIAL: NCT05452408
Title: PK Analysis of Antitumor B KAC in Patients with Oral Cancer
Brief Title: Antitumor-B KAC PK Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study abandoned.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Stuart Wong, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-WONG-ATB-KAC
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity
Keywords: Antitumor B KAC; Antitumor B Key Active Components
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Antitumor B KAC (Experimental): ATB will be administered on an outpatient basis.
  Interventions: Drug: Antitumor B KAC

INTERVENTIONS:
Drug: Antitumor B KAC — ATB-KAC will be administered at a dose of 720 mg three times per day (roughly spaced every eight hours) as has been studied for ATB-KAC in human oral leukoplakia trials and in esophageal cancer prevention trials. ATB-KAC may be taken with or without food.

SUMMARY:
Study Design: A Window of Opportunity Clinical Trial. This study design permits examination of effects of an oral agent on cancer patients during the "window" between diagnosis of their cancer and their definitive cancer surgery. Similar to a phase 0 study, the trial design permits examination of the biologic effects of an agent; in this study pharmacokinetic properties will be examined.

DETAILED DESCRIPTION:
Study Rationale: Establishing the PK profile for antitumor B key active components (ATB-KAC) is a critical initial step before future clinical trials can be performed that examine anticancer and cancer preventive effects of ATB-KAC.

Study Intervention Description: Study participants will take the natural botanical compound ATB-KAC during a short window (seven to 28 days). Participants will provide blood samples and saliva samples during ATB-KAC administration and a portion of the initial tumor biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of oral cavity squamous cell cancer.
2. Patient can start study agent administration but histological confirmation of squamous cell cancer (SCC) of the oral cavity (or histologic variants of SCC) by the pathologist must happen within seven days of registration in order to continue study agent administration.
3. Clinical stage II-IVA (as defined by the AJCC, 8th Edition) and amenable to surgical resection.
4. New diagnosis of oral SCC, new second primary, or recurrent oral SCC following a minimum remission of six months following previous definite surgery.
5. History and physical examination by an otolaryngologist and medical oncologist within 30 calendar days of study registration.
6. Study agent administration should start within seven days of registration.
7. Patient must receive administration of study agent for a minimum of seven days.
8. ECOG Performance status < 2.
9. Age ≥ 18 years.
10. CBC/differential obtained within 30 calendar days prior to registration, with adequate bone marrow function defined as follows:

    Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3; Platelets ≥ 100,000 cells/mm3; Hemoglobin ≥ 8.0 g/dL (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dL is acceptable.);
11. Adequate renal and hepatic function within 30 calendar days prior to registration, defined as follows:

    Serum creatinine < 1.5 mg/dL or creatinine clearance (CrCl) ≥ 50 mL/min within 14 calendar days prior to registration, determined by 24-hour collection or estimated by Cockcroft-Gault formula:

    CrCl male = [(140 - age) x (weight in kg)], [(Serum Cr mg/dL) x (72)] CrCl female = 0.85 x (CrCl male)
12. Total bilirubin < 2 x the institutional ULN within 30 calendar days prior to registration.
13. AST or ALT ≤ 3 x the institutional ULN within 30 calendar days prior to registration.
14. Glucose, potassium, and sodium within 30 calendar days prior to registration, with the following required parameters:

    Glucose: > 40 mg/dL or < 250 mg/dL; Potassium: > 3 mmol/L or < 6 mmol/L; Sodium: > 130 mmol/L or < 155 mmol/L.
15. Female patients must meet one of the following:

    * Postmenopausal for at least one year before the screening visit, or
    * Surgically sterile (i.e., undergone a hysterectomy or bilateral oophorectomy), or
    * If subject is of childbearing potential (defined as not satisfying either of the above two criteria), agree to practice two acceptable methods of contraception (combination methods requires use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 90 days after the last dose of study agent, AND o Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptom-thermal, post ovulation methods] and withdrawal are not acceptable contraception methods.)
16. Male patients, even if surgically sterilized (i.e., status postvasectomy), must agree to one of the following:

    * Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR
    * Must also adhere to the guidelines of any study-specific pregnancy prevention program, if applicable, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptom-thermal, post ovulation methods] and withdrawal are not acceptable methods of contraception.)
17. Patients must be deemed able to comply with the study plan.
18. Gastric tube study agent administration is permissible.
19. Patients must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

1. History of active liver disease.
2. Pregnant or lactating women are ineligible due to unforeseeable risks to embryo or fetus.
3. Concurrent use of any medicinal botanical, natural, or other herbal compound/s that the study PI believes could potentially have an impact on the results/objectives of this study.
4. Planned subtotal or debulking surgery, as determined by enrolling physician determination, is not permissible.
5. Prior systemic chemotherapy for oral SCC; note that prior chemotherapy for a different cancer is allowable.
6. Prior radiotherapy for oral SCC is permissible if disease free for one year since prior oral cancer treatment and free of significant late radiation effects.
7. Severe active comorbidity, such as uncontrolled cardiac disease, infection, severe COPD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Area under the Curve (AUC) for Saliva | predose, 30, 60, 120, 180, 240, 360, 480, and 1,440 min on Day 1
  The AUC will be calculated. The calculation will be mg/ml X hour.
Area under the Curve for Plasma | predose, 30, 60, 120, 180, 240, 360, 480, and 1,440 min on Day 1
  The AUC will be calculated. The calculation will be mg/ml X hour.
Cmax for Saliva | Day 1
  The Cmax will be calculated. The calculation will be ng/ml.
Cmax for Plasma | Day 1
  The Cmax will be calculated. The calculation will be ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J. Wong, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No